CLINICAL TRIAL: NCT00821951
Title: A Dose Escalation Study of Vorinostat in Combination With Palliative Radiotherapy for Patients With Non-Small Cell Lung Cancer
Brief Title: Vorinostat in Combination With Palliative Radiotherapy for Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0811004507
Record Dates: First submitted 2009-01-08; First posted 2009-01-14 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vorinostat; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vorinostat and Radiotherapy (Experimental)
  Interventions: Drug: Vorinostat; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Vorinostat — 200 mg, 300 mg, 400 mg, once per RT fraction
  Other Names: SAHA; Hystone Deacetylase (HDAC) inhibitor; ZOLINZA
Radiation: Radiotherapy — Standard fractionation of 3.0 Gy per day over 2 weeks, to a total dose of 30 Gy, will be utilized for all patients. All patients will be treated one time per day, 5 days per week unless interruption is clinically indicated.

SUMMARY:
This is a dose escalation study that will assess the safety of Vorinostat, a Histone Deacetylase (HDAC) inhibitor, in combination with palliative radiotherapy in patients with advanced or metastatic Non-Small Cell Lung Cancer (NSCLC). Vorinostat has been approved for use in patients with cutaneous T-cell lymphomas, but several pre-clinical studies suggest activity in lung cancer cell lines. Several HDAC inhibitors,including Vorinostat, may enhance the effect of radiotherapy, and this study will seek to confirm this.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility Criteria
* Patients must have histologically or cytologically confirmed NSCLC. Patients must have metastatic disease, stage IIIB with malignant pleural effusion, or be otherwise unsuitable for potentially curative therapy due to bulk of disease or comorbid medical illness. There must be disease apparent on imaging which offers a medical indication for radiation therapy. Palliative radiotherapy would be offered as appropriate standard therapy outside of a study setting. (NOTE: Radiotherapy utilized in this regimen is the same as that which would be offered as standard treatment outside of this study). Indications for palliative radiation include pain, pathologic fracture or risk of fracture, lymphovascular obstruction, bronchial obstruction, neural impingement, dyspnea, or bleeding.
* There must be a measurable tumor target (visible, palpable, or radiographically evident) for palliative radiation. The target for radiotherapy must be in the thoracic region (i.e., there must be normal lung tissue at the same anatomic level).
* Previous systemic therapy for NSCLC is allowed, as long as all prior therapy was completed at least two weeks before enrollment. Patients treated with nitrosurea or radioisotope may not be enrolled unless such treatment was at least 6 weeks prior to enrollment. Patients must have no previous exposed to HDAC inhibitors (patients previously treated with valproic acid are eligible if the exposure was greater than 30 days prior to enrollment).
* Age ≥18 years. Because no dosing or adverse event data are currently available on the use of vorinostat alone, or in combination radiation in patients <18 years of age, children are excluded from this study.
* ECOG performance status ≤3
* Life expectancy of greater 3 months.
* Patients must have normal organ and marrow function as defined below, all laboratory values to be obtained within 2 weeks prior to enrollment:
* absolute neutrophil count ≥1,500/mcL
* platelets ≥100,000/mcL
* hemoglobin ≥9 g/ dL
* serum bilirubin <1.5 times the upper limit of normal (ULN) serum AST, ALT, ALP <2.5 times ULN
* serum Creatinine <1.5 times ULN
* serum Potassium, Magnesium, Calcium - within normal range
* The effects of radiation on the developing human fetus are known to be teratogenic. For this reason, women of child-bearing potential and sexually active men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow a capsule
* Patients must have had a CT scan of the chest, abdomen, and pelvis (or PET/CT of the body), as well as an MRI or contrasted CT of the brain within 30 days of enrollment

Exclusion Criteria:

* Patients with known, untreated brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients who have received whole brain radiotherapy within 2 weeks of enrollment will also be excluded.
* Patients treated on an investigational drug trial within 30 days of study enrollment.
* Patients with active grade 2 or greater acute toxicity related to prior cancer-directed therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to vorinostat, or patients with a history of an unanticipated severe normal tissue reaction to previous radiation treatment.
* Patients with congenital long QT-syndrome will be excluded, as a known side effect of vorinostat is prolongation of QT interval. Patients on anti-arrhythmic medications or other medications known to lead to prolonged QT interval will be exclude unless an ECG has been obtained documenting a normal QT interval within 90 days prior to enrollment.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection (fever >38ºC within 48 hours of enrollment), symptomatic congestive heart failure (i.e., NYHA class 3 or greater), unstable angina pectoris, coronary angioplasty within 6 months prior to enrollment, or cardiac arrhythmia. Additionally, patients with suspected or confirmed poor compliance, mental instability, or prior or current alcohol or drug abuse deemed by the investigator to be likely to affect their ability to sign the informed consent, or undergo study procedures will be excluded.
* Pregnant women are excluded from this study because radiation has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with vorinostat, breastfeeding should be discontinued if the mother is treated. Women of childbearing potential must have a negative pregnancy test prior to enrollment.
* Patients with active HIV or viral hepatitis.
* Patients in whom primary radiation therapy, with potentially curative intent, is indicated will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-05; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Decker, M.D., Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients at Yale New Haven Hospital were recruited for a dose escalation trial between 2009 and 2010. Eligibility criteria included a histologic diagnosis of NSCLC, and an indication for palliative thoracic radiation in patients with either metastatic disease or locally advanced disease that precluded potentially curative therapy.
Pre-assignment Details: ECOG PS of 0 to 2, and adequate hematologic, hepatic, and renal function were required. Patients with prolonged QT syndrome or significant cardiovascular disease were excluded, as were patients with untreated brain metastases. Prior thoracic radiation was permitted as long as a treatment field could be designed without significant overlap
Groups:
- Vorinostat and Radiotherapy: Vorinostat : 200 mg, 300 mg, 400 mg, once per RT fraction
  Radiotherapy : Standard fractionation of 3.0 Gy per day over 2 weeks, to a total dose of 30 Gy, will be utilized for all patients. All patients will be treated one time per day, 5 days per week unless interruption is clinically indicated.
Period: Overall Study
Arm/Group | Vorinostat and Radiotherapy
Started | 17
Completed | 12
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Vorinostat and Radiotherapy
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of the Study is to Establish the Maximum Tolerated Dose of Vorinostat When Given Concurrently With Palliative Radiation.
Description: maximum tolerated dose of vorinostat when given concurrently with radiation
Time Frame: 1 Year
Population: All participants who received any drug
Measure: Number; unit: mg
Arm/Group | Vorinostat and Radiotherapy
Number analyzed (Participants) | 16
mg | 400

2. Secondary Outcome: Target Lesion Response
Time Frame: 1 Year
Reporting Status: Not Posted

3. Secondary Outcome: Vorinostat Modification of the DNA Damage Response in Patient Samples
Time Frame: 1 Year
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Vorinostat and Radiotherapy
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 8/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vorinostat and Radiotherapy (N=16)
hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
fatigue (General disorders) | 2 (2)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes